CLINICAL TRIAL: NCT04895098
Title: Retrospective Observational Study of the Efficacy and Safety of Statin Monotherapy or Statins in Combination With Ezetimibe in Patients Receiving Lipid-lowering Therapy in Both Primary and Secondary Prevention of CVD
Brief Title: Statin Monotherapy or Statins in Combination With Ezetimibe in Patients for Prevention of CVD
Acronym: UNISON
Status: Completed | Type: Observational
Sponsor: Akrikhin (Industry)
Collaborators: Russian National Atherosclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: EZE-01/21
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Lipid Metabolism Disorders; Cardiovascular Diseases
Keywords: Ezetimibе; Statin; Cardiovascular diseases; Lipid-lowering therapy
MeSH Terms: conditions — Lipid Metabolism Disorders; Cardiovascular Diseases | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- combination therapy group: 750 Subjects in the statin and ezetimibe combination therapy group
  Interventions: Drug: statin and ezetimibe combination therapy
- monotherapy group: 250 Subjects in the statin monotherapy group
  Interventions: Drug: statin monotherapy

INTERVENTIONS:
Drug: statin and ezetimibe combination therapy — Receiving statins (atorvastatin/rosuvastatin or others) in combination with ezetimibe 10mg/day in a stable dosing regimen (without changing the dose of the therapy and/or replacing the statin) for 3 or more months at the time of enrolment in the study.
  Other Names: no other intervention
  Groups: combination therapy group
Drug: statin monotherapy — Receiving statins (atorvastatin/rosuvastatin or others) as monotherapy in a stable dosing regimen (without changing the dose of the therapy and/or replacing the statin) for 3 or more months at the time of enrolment in the study.
  Other Names: no other intervention
  Groups: monotherapy group

SUMMARY:
Retrospective observational study of the efficacy and safety of statin monotherapy or statins in combination with ezetimibe in patients receiving lipid-lowering therapy in both primary and secondary prevention of cardiovascular diseases (CVD). The study will include patients receiving lipid-lowering therapy in both primary and secondary prevention of CVD who have received therapy of interest for ≥ 3 months in the 2 years preceding the signing of informed consent, i.e. statins as monotherapy or in combination with ezetimibe in a stable mode (without dose adjustment and/or statin replacement). Effectiveness of therapy will be evaluated based on the data on changes in baseline levels of total cholesterol (CS), low density lipoproteins (LDL), high density lipoproteins (HDL), triglycerides (TG), data on which will be obtained from primary medical records. Demographic and anthropometric data on patients, information on the history of hyperlipidemia and concomitant diseases will also be obtained. Also, the study will collect data on the development of adverse reactions of particular interest during therapy (liver/muscle damage, major cardiovascular events (MACE).

ELIGIBILITY:
Inclusion Criteria:

Patient can be included in the study only once.

1. Age > 18 years.
2. Patient receiving lipid-lowering therapy with statin monotherapy or statins in combination with ezetimibe for both primary and secondary prevention of CVD.
3. Receiving statins as monotherapy or statins in combination with ezetimibe in a stable dosing regimen for 3 or more months at the time of enrolment in the study.
4. Willingness and ability to sign an informed consent to participate in the study.
5. Availability of primary medical documentation, which allows assessment of all parameters necessary for the study from the moment of initiation of statin monotherapy or statins in combination with ezetimibe.
6. Initiation of lipid-lowering therapy not earlier than 2 years before enrolment into the study.

Exclusion Criteria:

1. Age < 18 years.
2. A diagnosis of familial hypercholesterolemia made prior to study enrolment or the investigator's suspicious of the possible presence of familial hypercholesterolemia.
3. Change in lipid-lowering therapy within 3 months prior to study enrolment.
4. Concomitant administration of omega-3 PUFA with statin monotherapy or combination therapy of statins and ezetimibe, as well as the use of any methods of extracorporeal filtration and/or plasmapheresis.
5. Clinically significant impairment of liver and/or kidney function, which may impede interpretation of test results
6. Presence of hypothyroidism
7. Ezetimibe monotherapy
8. Intolerance to statins at any dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients receiving lipid-lowering therapy in both primary and secondary prevention of CVD who have received therapy of interest for ≥ 3 months in the 2 years preceding the signing of informed consent, i.e. statins as monotherapy or in combination with ezetimibe in a stable mode (without dose adjustment and/or statin replacement).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Frequency of achieving target LDL (%) | at the time of enrolment in the study
  Frequency of achieving target LDL cholesterol levels at the time of enrolment (%)
Average change in LDL (absolute difference) | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Average change in LDL cholesterol level from the moment of the index event to inclusion (absolute difference)
Average change in LDL (% from the baseline) | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Average change in LDL cholesterol level from the moment of the index event to inclusion (% from the baseline)
Average change in total cholesterol (% and absolute difference) | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Average change in total cholesterol level from the moment of the index event to inclusion (% and absolute difference)
Average change in LDL (% and absolute difference) | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Average change in LDL cholesterol level from the moment of the index event to inclusion (% and absolute difference)
Average change in TG (% and absolute difference) | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Average change in TG level from the moment of the index event to inclusion (% and absolute difference)
The incidence of liver damage | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  an increase in ALT/AST levels over 1.5 of the upper limit normal [ULN]
The frequency of development of muscle damage | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  an increase in CPK level while excluding other possible factors of the development of the disorder
Major adverse cardiovascular events (MACE) incidence | from the moment of initiation of lipid-lowering drug therapy (not earlier than 2 years before enrolment into the study) to inclusion in the study
  Within the framework of this study, major adverse cardiovascular events (MACE) are considered as follows: myocardial infarction (MI), unstable angina pectoris, ischaemic stroke, aortocoronary bypass, mammary coronary bypass, coronary artery bypass, peripheral artery surgery, atherosclerotic stenosis of any artery more than 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Igor V Sergienko, MD,PHD,Prof., Principal Investigator — Russian National Atherosclerosis Society
Locations (31):
- Russia (31):
  - FGBOU VO "ChGU named after I.N. Ulianova", Cheboksary
  - FGBOU VO "ChGMA" Ministery of Health Russia, Chita
  - Gbuz "Iokb", Irkutsk
  - Gauz "Gkb #7", Kazan'
  - Nii "Kpssz", Kemerovo
  - KOGBUZ "Severnaya klinicheskaya bolnitca skoroi meditcinskoi pomotschi", Kirov
  - OOO TsEN YUG, Krasnodar
  - GUZ "Lipetskaya Gorpolyklinika #7", Lipetsk
  - ООО "MC "Semeiny doctor", Magnitogorsk
  - OOO "Semeiny doctor", Magnitogorsk
  - Fgbu Mnic Pm Ministry of Health Russia, Moscow
  - OOO ''Ne bolit", Moscow
  - FGBU NMIC of Cardiology Ministry of heath RF, Moscow
  - FGBOU DPO RMANPO Ministry of Health, Moscow
  - Chuz ''Ckb Rzhd Medicina", Moscow
  - Osp Rgnkc, Moscow
  - GBUZ NO "Gorodskaya Klinicheskaya Bolnitsa #38", Nizhny Novgorod
  - Gbuz No "Gkb #5", Nizhny Novgorod
  - OOO "DaVinchi-NN", Nizhny Novgorod
  - NII TPM - affiliate of SO RAN, Novosibirsk
  - Buzoo "Kkd", Omsk
  - Gbus "Bsmp", Petrozavodsk
  - FGBOU VO SZGMU named after I.I.Mechnikov, Saint Petersburg
  - FGBU "SZONKC named after L.G.Sokolov FMBA of Russia", Saint Petersburg
  - Ooo "Veraks-Med", Saint Petersburg
  - GBUZ "SOKKD named after V.P.Polyakov", Samara
  - Fgbou Vo Tyumensky Gmu Ministry of Health Russia, Tyumen
  - Cardiology cabinet "Serdce pod zaschitoy" IP Barov P.A., Ulyanovsk
  - GBUZ VO "City hospital #4 of Vladimir", Vladimir
  - GBUZ VO "GB #4 c. Vladimir", Vladimir
  - FGBOU VO "UGMU" Ministry of Health Russia, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No